CLINICAL TRIAL: NCT06647342
Title: Randomised Controlled Clinical Trial Investigating the Effect of Reduced Bleomycin in Elechtrochemotherapy Treatment on Patients With Cutaneous Malignancies (The BLESS Trial)
Brief Title: The Effect of Reduced Bleomycin in Electrochemotherapy Treatment
Acronym: BLESS
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Julie Gehl (Other)
Collaborators: Roskilde University (Other); Herlev Hospital (Other)
Responsible Party: Sponsor-Investigator, Julie Gehl, Professor, Zealand University Hospital
Organization: Zealand University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CTIS: 2024-513360-25-00; 2024-513360-25-00 (EU CTIS Number)
Record Dates: First submitted 2024-10-13; First posted 2024-10-17 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2024-10

CONDITIONS: Cutaneous Metastasis; Cutaneous Malignant Mixed Tumor; Bleomycin Adverse Reaction; Electrochemotherapy
Keywords: Deescalating study; Bleomycin; Electrochemotherapy; Cutaneous malignancies; Cutaneous tumors
MeSH Terms: conditions — Skin Neoplasms | interventions — Bleomycin

STUDY DESIGN:
Intervention Model Description: Double-blinded randomized controlled study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Investigators analysing bleomycin concentrations using HPLC.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Standard dose (Active Comparator): Patients in this arm will recieve the standard dose of bleomycin during treatment with electrochemotherapy
  Interventions: Drug: Bleomycin
- Dose reduction (Experimental): Patients in this arm will recieve half the standard dose of bleomycin during treatment with electrochemotherapy
  Interventions: Drug: Bleomycin

INTERVENTIONS:
Drug: Bleomycin — In the standard arm, Bleomycin (Baxter, Germany) at a dose of 15.000 IU/m² is used. In the dose reduction arm, a dose of 7500 IU/m² is used. Note that in Denmark bleomycin is dosed by international units, whereas other countries may use respectively U (units) or mg.

SUMMARY:
The objective of this trial is to determine if reducing the chemotherapy dose in electrochemotherapy is equally effective as using the standard dose for treating various types of skin tumors.

Electrochemotherapy involves administrating chemotherapy intravenously, followed shortly by a brief electrical pulse to the tumor. This pulses temporarily increases the tumor cells permeability, allowing the chemotherapy to enter more effectively.

Participants will undergo a single session of electrochemotherapy with either half the standard chemotherapy dose or the full standard dose. The size of the cutaneous tumors will be measured before treatment and again three months after the treatment to compare their response in both groups. To monitor the tumors, as well as assess the adverse events and quality of life, participants must attend follow-up visits at two weeks, three months and twelve months. Additional visits may be scheduled at one, two, four and six months, if necessary, as determined by the clinician or the patient. Concentration of chemotherapy will be measured in blood samples and in samples from the treated tumor and normal skin.

DETAILED DESCRIPTION:
Introduction

Electroporation Electroporation is a method in which the cell is exposed to an external electric field resulting in increased permeability of the cell membrane [1]. Electroporation is used to introduce drugs into cells, without affecting intracellular organelles or cell viability. By inducing this response, drugs that are normally non-permeant, e.g. hydrophilic chemotherapy such as bleomycin, will enter the cell by diffusion thus enhancing the cytotoxic effect [2, 3]. The combination of electroporation and chemotherapy is known as electrochemotherapy (ECT). The application of the electric pulses causes vasoconstriction, inducing drug entrapment due to reduced blood flow - this is termed the vascular lock [4, 5]. In addition, electroporation also has a vascular-disrupting effect, when combined with chemotherapy [4]. ECT damages tumour vasculature leading to an additional cascade of tumour cell death due to lack of oxygen, nutrients, and waste product accumulation [5]. These vascular changes are more prolonged in tumours than in normal tissue [6].

Electrochemotherapy ECT is the combination of chemotherapy and electroporation, in which electric pulses are administered to a tumour after intravenous or intratumoural injection of chemotherapy. ECT has been shown to be effective in the treatment of cutaneous malignancies and is established as standard treatment for cutaneous primary and secondary skin tumours and ulcerating malignant wounds [7, 8]. ECT is often used as a one time treatment, but can be repeated if necessary.

Bleomycin is the drug of choice for ECT; it has low toxicity to normal cells and the largest increase in efficacy after electroporation enhancing the cytotoxic effect with a factor 300 to 5.000 [9]. ECT is performed in general or local anaesthesia depending on tumour location and size. Patient preference and institutional practice is also taken into account [8].

Bleomycin is an antineoplastic drug derived from Streptomyces verticillus and is used in the treatment of a variety of malignancies, such as lymphoma and testicular cancer [11]. Bleomycin generates single- and double-strand DNA breaks, i.e., one molecule of bleomycin can cause 10-15 DNA strand breaks [12]. Due to its hydrophilic nature, the entry of bleomycin into cells is restricted and occurs via an endocytotic process [13]. Bleomycin causes cell death in two ways, depending on the doses used: 1) if a lower amount of bleomycin is used (thousands of bleomycin molecules) the cell arrests in the G2-M phase, enlarges and becomes polynucleated and dies slowly by necrosis; 2) if a larger amount is used (millions of bleomycin molecules), pseudo-apoptosis kills the cell within a few minutes [12, 14].

Recently, it has been shown that the disaccharide moiety of bleomycin facilitates uptake by cancer cells. It is suggested that the upregulation of receptors associated with enhanced glycolysis in tumour cells could be the reason for bleomycin targeting tumour cells selectively [51].

Bleomycin is degraded by an enzyme - bleomycin hydrolase -, found in various normal tissues [11]. A lower concentration of this enzyme is found in the skin and lungs, which can lead to increased harms in these organs [15, 16]. The Danish Medicines Agency (DMA) states in its product summary that half of patients receiving bleomycin experience harms related to the skin (erythema, hyperpigmentation, striae or soreness) and one tenth experience pulmonary reactions with a minority (1%) dying from pulmonary fibrosis [15]. Some studies have observed that the risk of developing pulmonary toxicity from bleomycin is increased with age, drug dose, and concomitant oxygen therapy and thoracic radiation therapy [16].

Since harms are associated with accumulative bleomycin dose, it is desirable to investigate if the dose can be reduced to minimize risk of harms and maintain the same efficacy. This may also enable some ineligible fragile patients to become eligible for ECT treatment, e.g., lung cancer patients with a higher risk of developing pulmonary toxicity.

Cutaneous malignancies A significant proportion of cancer patients develop cutaneous metastases (~10%) that often become exuding, bleeding or odorous [17, 18]. Thus, the metastases may influence patients' quality of life [19, 49]. Cutaneous metastases negatively affect patients, i.e., self-esteem, body image, and sexuality with feelings tied to frustration and loss of power [21, 22]. Most cancer patients receive chemotherapy or immunotherapy, but some cancers do not respond to these standard treatments [23]. ECT may be used for such cancers enhancing palliation and quality of life [3, 24]. The most frequently seen cutaneous metastases originate from breast cancer and occur in the chest region, but may arise anywhere on the body and originate from most cancer types [20]. The cutaneous malignancies may vary in size from a few millimetres to very large and may be focal or extensive.

Clinical experience with electrochemotherapy In 1993, Belehradek and colleagues published the first clinical trial of ECT using bleomycin in 8 patients indicating that the treatment was well-tolerated by patients and with a clinical complete rumour response of 57% [25]. In 2003 Gothelf and colleagues reviewed the 11 clinical trials completed between 1993 and 2001, involving a total of 96 patients with 411 tumours/metastases treated with different approaches [26]. The overall response (OR) varied between 15% and 100%. For the 11 ECT studies investigating bleomycin and ECT treatment on cutaneous malignancies the OR has been between 22% and 100%. Three studies stand out, with an OR of 22%, 28% and 45%, respectively [27-29]. The study by Domenge from 1996, was one of the first studies conducted on ECT and included only seven patients [27]. In the studies by Matthiessen and Kreuter larger tumours (>3 cm) were included. It is well-known that the size of the tumour affects the response of the ECT treatment [29]. When excluding these studies the OR varies from 58% to 100%. The largest ECT bleomycin study by Clover and colleagues from 2020 included 987 patients with 2,483 tumours [30] and showed that different tumours have different ORs; for example, basal cell carcinoma (BCC) and Kaposi's sarcoma (KS) show the highest OR with 96% and 98%, respectively; while breast cancer metastases, malignant melanoma (MM) and squamous cell carcinoma (SCC) have lower responses of 77%, 82% and 80%, respectively. This study also observed an effect of tumour size on the overall tumour response. The highest response rates were observed in small tumours (<3 cm). In small skin metastases (<2 cm), no significant OR difference was observed between intravenous vs. intratumoural administration of bleomycin, however, for larger skin metastases (>2cm), the OR was significantly (p<0.05) higher with intravenous administration (57% vs. 48%) [30]. Thus, our trial will be stratified according to tumour/metastasis size.

Clinical experience with reduced bleomycin In 1996, one of the first clinical ECT bleomycin studies with six patients used a bleomycin dose of 10.000 IU/m2 [31] (see Table 1), since medical and surgical oncologists believed that a dose of 22,700 IU/m2 - used in the first clinical trials - was too high. This is the only study using this dose and from 1998 the standard dose of 15.000 IU/m2 was used in most studies.

In 2016, a case report of a patient receiving ECT with bleomycin with a 50% reduced dose (7.500 IU/m2) due to renal dysfunction was published. In this case a complete tumour response was observed [32].

From 2013 to 2016, Rotunno identified via the International Network for Sharing Practices on Electrochemotherapy (InspECT) database 57 patients treated with ECT and reduced bleomycin (7.500, 10.000 or 13.500 IU/m2) [33] due to e.g., reduced renal function and high age. Reduced bleomycin showed similar tumour response to a standard bleomycin dose (15.000 IU/m2), with an OR of 64% to 82 %. Thus, the authors of the study suggested that reduced bleomycin doses could be as effective as the standard treatment - especially in patients with impaired renal function or patients eligible to multiple ECT cycles. It was concluded that further research in order to find a personalized bleomycin dose is needed [33].

In 2018 and 2021, two studies concluded that a reduced dose of bleomycin is a feasible treatment option for elderly patients, with equal efficacy to standard dose treatment (OR 87% to 100%) and should be considered as a treatment in patients with comorbidities [34, 35]. In addition, in a study by Groselj et al. from 2018 it was suggested that the cosmetic outcome was improved with the use of a reduced dose of bleomycin compared to the standard dose due to shorter healing and less development of fibrous scarring tissue [36].

Rationale for 50% bleomycin reduction in this study:

Based on former literature [32-36] we find it realistic to reduce the bleomycin dose with 50% and still gain a sufficient overall tumour response after ECT treatment. For time efficiency purposes, in this study we have decided to investigate a 50% reduced dose of bleomycin only. Randomisation to several bleomycin dose levels would subsequently result in the need of a significant increase in the number of included patients and/or referring hospital departments, which would be time consuming and difficult to complete within a manageable time frame.

Methods Trial design The study design as a non-inferiority study and is a parallel two-armed double-blinded randomized clinical trial, where the patients are stratified due to the size of their biggest cutaneous tumour (≤ 3 cm or > 3 cm) and afterwards randomized (1:1) to receive a standard dose bleomycin or a 50% reduced dose bleomycin.

Blinding is performed by the pharmacy mixing the allotted dose regimen after randomization, both patients and treating staff will be blinded to the bleomycin dose. Unblinding will be performed according to procedure if need be. Unblinding of all results will take place after last patients evaluation of primary endpoint.

The study will be conducted at two centers in Denmark: At the department of Clinical Oncology and Palliative Care, Zealand University Hospital, Roskilde and at the Department of Oncology, Copenhagen University Hospital, Herlev Gentofte Hospital. The three year study period is expected to start in October 2024.

Study population Patients will be referred from oncologic departments and must be advised about treatment alternatives. It must be evaluated whether the patient will benefit from the treatment, given the localisation and size of the tumour/tumours, the patient's general condition and expected survival. The purpose, possible risks and benefits should be discussed in collaboration with the patient.

Indications for participating in this trial includes:

* Biopsy verified cutaneous malignancies of any histology, which are symptomatic due to bleeding, ulceration, oozing, odour, or pain
* Primary skin cancers, including recurrent tumours, where other treatment modalities have failed, are not possible or not appropriate
* Patients who are receiving systematic anti-neoplastic therapy, but where cutaneous metastases are progressing or not responding despite satisfactory response to systemic therapy in internal organs
* Patient preference for electrochemotherapy, after other treatment possibilities have been thoroughly explained to the patient For eligibility criteria, please refer to the section about eligibility criteria.

Pre-treatment examination and pain management:

The pre-treatment examination will be performed up to one month prior to the procedure and will include diagnosis of primary tumour, TNM (tumour, node, and metastasis) classification, and previous anti-neoplastic treatments. Under previous treatments, it must be noted which nodules have been treated with which treatment. Radiotherapy fields or other local treatments must be listed if nodules were subjected to this. Additionally, assessment of medical history, previous problems with anaesthesia, any other relevant medical history, combination with other treatments, and presence of symptoms will be noted. A physical examination with clinical assessment of the tumour, location and availability of electroporation will be made. All the cutaneous tumours of the patient will be treated, but a maximum of seven tumours per patient will be registered and followed over time, and only one tumour will be selected for tissue biopsies.

Moreover assessment of performance status will be performed, and pre-existing pain problems will be examined in order to create a pain management plan.

Treatment day Anaesthesia As this is a study including treatment with intravenous bleomycin, participants will in most cases receive general anaesthesia, administered according to institutional guidelines or standard operating procedures [52]. In cases where local anaesthetics are preferable, this can also be utilized and administered according to institutional guidelines.

Bleomycin dose Bleomycin is the approved chemotherapeutic drug for use in ECT and will be used according to the marketing authorization in this trial.

In order to calculate the body surface area (BSA), the patients' height will be noted and their weight measured. Patients will receive either a standard dose of bleomycin (15.000 IU/m2 BSA) or a dose reduced with 50% (7.500 IU/m2 BSA) intravenously. Bleomycin is infused over a short time (2-5 min) and 8 min after completion of the infusion, the drug has diffused into tumour tissues and hereafter the electric pulses can be applied.

Applied electric pulses The electric pulses will be administered 8 minutes after bleomycin infusion. It is important that the entire tumour volume with surrounding tissue is treated with electroporation, so a margin of 3 mm around the tumour is included in the treatment.

For electroporation we use the Cliniporator (model EPS02, IGEA, Carpi, Italy), square wave pulse generator, which delivers a series of eight consecutive pulses of 0.1 msec each with an amplitude of 1 kV/cm and a frequency of 1 Hz. The electrodes will be chosen according to the standard operating procedures [8], depending on size and anatomical location of the tumour.

All tumours will be treated, but a maximum of seven tumours per patient will be followed, and only one tumour will be selected for tissue biopsies.

Biological samples Two biopsies from normal skin surrounding the tumour will be collected: one before bleomycin infusion and one 8 minutes after bleomycin infusion. Five biopsies will be collected from each patient from one of the tumours, at the time points; before bleomycin infusion, 2, 4, 6 and 8 minutes after bleomycin infusion. An additional tumour biopsy will be collected before bleomycin infusion for histologic analysis, this biopsy will (optional to the patient) be repeated after one year. The biopsies will include 3 mm tissue per biopsy and a maximum of 0.75 ml.

Six blood samples will be collected at predetermined time points at treatment day (before bleomycin infusion, 5, 10, 20, 30 and 40 min after bleomycin administration.

The blood and biopsies (except those made for histological analysis) will be analysed at the Department of Science and Environment at Roskilde University according to the amount of bleomycin. Here the HPLC machine will be used to detect the All blood samples will be stored in a collective bio bank situated at Region Zealand Biobank approved by the Danish Data Protection Agency.

Follow up Mandatory follow-ups occur at 2 weeks, 3 months and 12 months. Optional follow-up consultations will be possible at 30, 60, 120 and 180 days after ECT treatment. The necessity of these optional consultations will be decided by the physician and patient.

Each target tumour size will be assessed with a ruler and documented with photography's before treatment and at all the follow up consultations. At 3 months and 12 months evaluation of wound healing and scar formation will be accessed by three independent observers (1 plastic surgeon, 1 oncologist, and 1 research associate) using the Vancouver Scar Scale and the Patient and Observer Scar Assessment Scale. Moreover quality of life EORTC-questionnaires will be performed. At all follow-up consultations pain from the tumours and adverse events will be measured.

For primary and secondary endpoints, please refer to the relevant sections.

Methods employed for evaluation of quality of life Patients will be asked to answer the European Organisation for Research and Treatment of Cancer (EORTC) QLQ-C30 questionnaire at month 0, 3 and 12. This questionnaire is developed to assess the quality of life of cancer patients.

Additionally, 16 patients will participate in a qualitative interview at baseline and at month 3 if they give separate consent. This is in order to learn about patient experiences with treatment and to assess ECT treatment impact on quality of life. In this study qualitative interviews may uncover concerns and priorities that distinguish cancer patients with cutaneous malignancies from other patients and thereby help to sufficiently capture the patient's experience [38]. To collect patient experiences, semi-structured interview is chosen as it gives the researcher the freedom to probe the interviewee to elaborate or to follow a new line of inquiry introduced by what the interviewee is saying.

Sample size:

This is a non-inferiority study, where the primary endpoint is to compare overall response at tumour level three months after ECT treatment with two different doses of bleomycin. The appropriate sample size is calculated to determine the minimum number of tumours that need to be treated in this study in order to have a sufficient statistical power showing that halving the dose of bleomycin is non-inferior to the standard dose.

To calculate the sample size, we utilized the formula for non-inferiority study with continuous data [37]. The standard deviation was derived from 55 studies from 1996 - 2021 exploring electrochometherapy with intravenous bleomycin in different tumour histologies [38]. We assumed an acceptable response rate difference on 10%. The significance level where set at 0.05 with 80% power. Based on the findings on five previous studies, where there was observed a drop-out rate at 16% [30, 39-42], we conservatively estimated a drop-out rate at 20%. This led to the conclusion that 110 tumours needed to be treated in this study. Anticipating an average of approximately 2 tumours per patient to be evaluated, as observed in previous literature [30], we plan to enroll 55 patients.

Recruitment Patients will be recruited from four departments: the Department of Clinical Oncology and Palliative Care and the Department of Plastic and Breast Surgery at Zealand University Hospital Roskilde, and Department of Oncology and Department of Plastic Surgery at Herlev Hospital, respectively. Patients eligible for treatment might be referred from other departments throughout Denmark.

End of Trial The trial will conclude when 55 patients have been enrolled, have received ECT, and the last patient has completed their final scheduled follow-up (12 months after ECT).

ELIGIBILITY:
Inclusion Criteria:

1. Trial subject > 18 years.
2. Trial subject must be able to understand the participant information.
3. Histologically verified cutaneous or subcutaneous, primary or secondary cancer of any histology.
4. Life expectancy > 3 months.
5. Trial subject can undergo simultaneous medical treatment (endocrine therapy, chemotherapy, immunotherapy, etc.) at any point during the study.
6. Trial subject may have received ECT treatment previously if selected tumours have not received ECT or if a minimum of 3 months after ECT treatment have passed.
7. Trial subject can undergo radiation therapy, provided that the treatment field does not involve the area intended to treat. If the trial subject has received radiation therapy in the area intended to treat, a minimum of 3 months should have passed.
8. A creatinine level within normal upper limit. If creatinine is above normal upper limit the subject needs to have a creatinine clearance > 50 ml/min.
9. Both men and women who are sexually active must use safe contraception. This includes the use of intrauterine device (IUD), oral contraceptives, male or female condom, vasectomy or female sterilization.
10. Signed informed consent.

Exclusion Criteria:

1. Pregnancy or lactation. All fertile women will have to deliver a negative pregnancy test before ECT treatment.
2. Allergy or hypersensitivity to bleomycin.
3. Acute lung infection.
4. Severely impaired lung function or any lung condition the investigator deems severe.
5. Any other caution, clinical disease or previous treatments that make the investigator deem the trial subject unfit.
6. The cumulative bleomycin dose must not exceed the by the drug manufacturer recommended maximum dose.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2024-10-29 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the clinical overall response rate of electrochemotherapy treatment of cutaneous malignancies after three months | The tumors will be meassured before electrochemotherapy (baseline) and three months after electrochemotherapy treatment.
  The response to treatment will be evaluated according to the modified Response Evaluation Criteria in Solid Tumours (RECIST) criteria. Response rate will be defined as the number of responding tumours relative to the number of treated tumours (Intention to treat analysis, ITT), evaluated 3 months after treatment. The response will be evaluated by clinical examination with ruler measurements (in mm) and photographical documentation using rulers for scale.

SECONDARY OUTCOMES:
Treatment response for normal dose group, reduced dose group, and for all treated tumors at optimnal time points using the mRECIST criteria. | The follow up is mandatory for the patients after 2 weeks, after 3 months and 12 months. Follow up is optional at 1 month, 2 moths, 4 moths and 6 months. At every visit the tumours size will be measured.
  Tumors size in mm are measured with a ruler and documented with digital photographies.
Aesthetic outcome for normal dose group, reduced dose group and for all tumours 3 months after treatment and 1 year after treatment, using the Vancouver Scar Scale. | Assessed 3 months after treatment and 1 year after treatment.
  The Vancouver Scar Scale assesses scars based on four criteria: vascularity, pigmentation, pliability and hight. Each scar or lesion is evaluated given a score ranging from 0 to 13, with 13 representing the most severe scar.
Aesthetic outcome for normal dose group, reduced dose group and for all tumors assessed at 3 month and 12 month, using Patient and Observer Scar Assessment Scale (POSAS). | 3 months ater treatment and 1 year after treatment.
  Patient and Observer Scar Assessment Scale (POSAS) is a tool used to evaluate scars both from the patient's and the observer's persepective. Each independently completes a questionnaire assessing various aspects of the scar, such as color, thickness, and overall appearance. All questions are rated from "not" to "extreamly", to capture the severety of each feature.
Complete and partial remissions for all patients treated (patient level) | Before treatment (baseline) compared to 3 months after treatment.
  Response at patient level defined as number of patients experiencing objective responses on at least one treated tumour.
Biopsy at 12 months (optional) for histological examination of malignancy presence (HE stain, and staining for specific tumour markers can be included). | 12 months
  Biopsy confirmation of response at 12 months.
All-cause mortality and cancer related mortality within 12 months. | Study period of 12 months.
  Mortalities during the study period will be registered and classified by cancer related mortality and all-cause mortality.
Quality of life before treatment and at approximately 3 months measured by EORTC-QLQ-C30 | Questionaires will be performed before electrochemotherapy, and at 3 and 12 months after the treatment. .
  The questionnaire consist of 28 questions regarding the patient and their health. For each question the patient selects one of four options: "not at all", "a little", "quite a bit" and "very much" when anwering the questions. At the end there are two additional questions, where the patient rates their overall health and quality of life during the past week.
Quality of life before treatment and 3 months post-treatment measured in 16 patients with semi-structured qualitative interviews. | Qualitative interviews will be performed before electrochemotherapy and 3 months post-treatment in the same patients.
  Qualitative interviews, optional to the patients and ideally conducted in 16 participants, will take place either in the patients' home or another location of their choice. Each interview will last for approximately an hour and will follow a semistructured interview-guide.
Relation between tumour histology and tumor response rates at 3 months and 12 months. | Response rate will be calculated by comparing measurement at baseline and at respectively 3 months, and at 12 months.
  Cutaneous metatases of different cancer histologies are treated in this protocol, and response rates will given by cancer histology (descriptive statistics). Response rate will be calculated for each tumor histology by comparing baseline measurements with response according to RECIST criteria, as respectively 3 and 12 months.
Response rates in tumours according to size | Baseline measurement will be compared to measurements at respectively 3 months and 12 months.
  Response rates will be investigated according to tumor size (up to 3 cm or over 3 cm).
Side effects according to CTCAE according to treatment dose - data from normal dose group, reduced dose group, and for the whole population will be registered and compared. | Will be meassured at every visit up to one year
The presence of pain (if any) associated with the cutaneous malignancies will be assessed using Numeric Rating Scale (NRS). | Will be meassured at every visit up to 12 months.
  The numeric rating scale lists 0 as no pain at all and 10 as the worst imaginable pain, the scale going from 0 to 10.
Bleomycin pharmakokinetics at electrochemotherapy procedure | Blood samples will be drawn before bleomycin infusion (time 0), and at 5, 10, 20, 30 and 40 minutes after bleomycin infusion.
  Bleomycin will be measured in blood samples via UHPLC-ESI-MS and the outcome will be in ng/ml.
Bleomycin pharmakokinetics related to dose group, age and body surface area | Samples will be drawn before bleomycin infusion (time 0), and at 5, 10, 20, 30 and 40 minutes after bleomycin infusion.
  Bleomycin will be measured via UHPLC-ESI-MS and the outsome will be in ng/ml. Results will be categorised by treatment group (standard dose bleomycin group vs reduced dose belomycin group. Results will also by related to patient age and body surface area.
Bleomycin pharmakokinetics realted to kidney function. | Serum creatinine will be measured before treatment. Samples for bleomycin pharmakokinetics will be measured in blood drawn before bleomycin infusion (time 0), and at 5, 10, 20, 30 and 40 minutes after bleomycin infusion.
  Bleomycin will be measured via UHPLC-ESI-MS and the outsome will be in ng/ml. Kidney function is assessed by pre-treatment serum creatinine. Pharmakokinetics will be compared to kidney function.
Bleomycin concentration in tumours over time | Biopsies from tumor will be obtained before bleomycin infusion (0 min), 2, 4, 6, and 8 min. after bleomycin infusion.
  Tumor koncentration of bleomycin will be examined to understand relation to bleomycin pharmakokinetics in the same patient, as well as changes in tumor bleomycin koncentration in the time immediately following bleomycin administration. Bleomycin concentration in tumour will be measured (UHPLC-ESI-MS) in ng/ml.
The fraction of tumour cells will be related to the bleomycin concentration in tumor. | Pretreatment biopsy from tumor, obtained on the day of treatment.
  The percentage of tumor cells in a pretreatment biopsy (optained the day of treatment) will be compared to the amount of bleomycin in the same tumor.

CONTACTS AND LOCATIONS:
Overall Officials: Julie Gehl, Professor, MD, Study Chair — Department of Oncology and Palliative Care, Zealand University Hospital, Denmark
Locations (2):
- Denmark (2):
  - Copenhagen University Hospital Herlev-Gentofte, Herlev
  - Zealand University Hospital, Roskilde

IPD SHARING:
Plan to Share IPD: Yes
Pseudoanonymized data from patients will be uploaded to the InspECT-database (International Network for Sharing Practices on Elechtrochemotherapy).
Supporting Information: Study Protocol, CSR
Time Frame: Study protocol will be immediately available, and a protocol article will be written.
Access Criteria: Information regarding study protocol will be directly available from the investigator. Results from the study will be published in a peer reviewed international journal. Pseudoanonymized data will be uploaded to the Inspect database, but not otherwise be made available.

REFERENCES:
- [Background] Bastrup FA, Vissing M, Gehl J. Electrochemotherapy for metastatic cutaneous melanoma. Acta Oncol. 2022 May;61(5):531-532. doi: 10.1080/0284186X.2022.2057199. Epub 2022 Apr 29. No abstract available. PMID 35484987